CLINICAL TRIAL: NCT00000111
Title: Intraoral Grafting of Ex Vivo Produced Oral Mucosal Composites
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00042-1620; M01RR000042 (NIH)
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-09

CONDITIONS: Mouth Diseases
Keywords: mouth mucosa; transplants
MeSH Terms: conditions — Mouth Diseases

INTERVENTIONS:
Procedure: Oral mucosal graft

SUMMARY:
The purpose of this study is to see if we can develop a good graft for oral mucosal tissue that is like the top of the mouth in a "test tube" that could be used successfully in humans. We have already done this successfully mice. The next step is to take a small piece of tissue from a human volunteer and see if we can grow a larger piece of tissue from it outside the human body and graft it back into the same person successfully. We expect that this technique will work. It has already been tried in patients with burns of the skin who have had similar procedures where the skin is grafted back to them. The significance of this research is that oral tissue taken from the top of the mouth or palate is in limited supply and leaves the patient with a painful and uncomfortable post surgery experience. If we are successful with our technique the patient will experience less pain and discomfort from the site that we are using to grow our tissue outside the body than if we had taken it from the top of the mouth or palate. In addition, by waiting longer periods to grow the patient's cells we can make larger pieces of oral tissue than we could have gotten directly from the patient's mouth. Patients who will participate in this study will need to require a soft tissue graft from the mouth to an area that needs additional attached or keratinized mucosa. This will most likely be either in preparation for patients who have or will have dental implants placed. Another subset of patients are those who need scar tissue released or the vestibule of their mouth (area that turns from the gums to the lip) released.

ELIGIBILITY:
Inclusion Criteria:

* Lack sufficient attached keratinized tissue at recipient surgical site in question

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult